CLINICAL TRIAL: NCT04061252
Title: A Phase 3, Placebo-Controlled, Double-Blind Comparative Study of KHK4827 With an Open-Label Extension in Subjects With Palmoplantar Pustulosis
Brief Title: A Study of KHK4827 in Subjects With Palmoplantar Pustulosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4827-009
Record Dates: First submitted 2019-07-16; First posted 2019-08-19 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2022-04

CONDITIONS: Palmoplantar Pustulosis
Keywords: Palmoplantar Pustulosis; brodalumab; KHK4827
MeSH Terms: conditions — Psoriasis | interventions — brodalumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KHK4827 210mg Q2W SC (Experimental)
  Interventions: Drug: KHK4827
- Placebo Q2W SC (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KHK4827 — brodalumab 210mg Q2W, SC
  Arms: KHK4827 210mg Q2W SC
Drug: Placebo — Q2W, SC
  Arms: Placebo Q2W SC

SUMMARY:
Evaluation of efficacy and safety of KHK4827 in Subjects with Palmoplantar Pustulosis

ELIGIBILITY:
Inclusion Criteria:

* Subject has had a diagnosis of palmoplantar pustulosis for at least 24 weeks as of the time of informed consent.
* Subject has a PPPASI total score ≥12 and a PPPASI severity score of pustules/vesicles on the palms or soles ≥2 both at the pre-examination and enrollment examination;
* Subject inadequately responded to any one or combination of the following therapies before informed consent: Topical corticosteroids, Topical vitamin D3, Phototherapy, Etretinate

Exclusion Criteria:

* Subject has a diagnosis of plaque psoriasis, pustular psoriasis, drug-induced palmoplantar pustulosis, or pompholyx;
* Subject has an improvement in PPPASI total score of ≥4 points during the screening period;
* Subject has a history or evidence of psychiatric disorder or alcohol/drug abuse that, in the opinion of the investigator or subinvestigator, may compromise the safety of the subject because of participation in the study or may interfere with assessments and procedures in the study or study completion;
* Subject has a past or current history of suicidal ideation (severity of 4 or 5) or any suicidal behavior at enrollment, as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS);
* Subject has severe depression with a PHQ-8 total score of ≥15 at enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2019-08-10 (Actual); Primary Completion 2021-08-11 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Palmoplantar Pustulosis Area and Severity Index (PPPASI) total score at Week 16 | Baseline, Week 16
  PPPASI is composed of subscores of erythema (E), pustules/vesicles (P), desquamation/scales (D) on the left (L) and right (R) palm (P) and sole (S) respectively. PPPASI is calculated by the following calculation formula.
  PPPASI=(E+P+D) Area*0.2 (RP)+(E+P+D) Area*0.2 (LP)+ (E+P+D) Area*0.3 (RS)+(E+P+D) Area*0.3 (LS).

SECONDARY OUTCOMES:
Change from baseline in Palmoplantar Pustulosis Severity Index (PPP-SI) total score at Week 16 | Baseline, Week 16
  (PPP-SI) total score at Week 16. PPP-SI assesses the severity of palmoplantar pustulosis skin lesions and response to therapy. Scores can range from 0 to 12, with higher scores indicating more severity.
The percentage of participants who achieved at least 50% improvement in PPPASI score from Baseline to Week 16 | Week 16
The percentage of participants who achieved at least 75% improvement in PPPASI score from Baseline to Week 16 | Week 16
The percentage of participants who achieved a Physician's Global Assessment(PGA) score of 0 or 1 at Week 16 | Week 16
Change from baseline in PPPASI total score at each assessment time point | Baseline, Week 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68
Change from baseline in PPP-SI total score at each assessment time point | Baseline, Week 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68
Change from baseline in Dermatology Life Quality Index (DLQI) score at each evaluation point | Baseline, Week 8, 16, 24, 32, 44, 56, 68
  The DLQI is a skin disease-specific scale that assesses the impact of skin symptoms on QOL during the past 7 days and consists of 10 questions relating to "symptoms and feelings", "daily activities", "leisure", "work and employment", "personal relationship", and "treatment". The DLQI produces a numeric score that can range from 0 to 30. Higher score indicates more severe disease.

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Takagi Dermatology clinic, Obihiro, Hokkaido
  - Sapporo Dermatology clinic, Sapporo, Hokkaido

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Okubo Y, Kobayashi S, Murakami M, Sano S, Kikuta N, Ouchi Y, Terui T. Efficacy and Safety of Brodalumab, an Anti-interleukin-17 Receptor A Monoclonal Antibody, for Palmoplantar Pustulosis: 16-Week Results of a Randomized Clinical Trial. Am J Clin Dermatol. 2024 Sep;25(5):837-847. doi: 10.1007/s40257-024-00876-x. Epub 2024 Jul 2. PMID 38954226